CLINICAL TRIAL: NCT07325565
Title: Impact of Emotional Disorders on Response to Immune Checkpoint Inhibitor Therapy in Liver Cancer: A Multicenter, Prospective, Multi-Cohort Study
Brief Title: Impact of Emotional Disorders on Response to Immune Checkpoint Inhibitor Therapy in Liver Cancer
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Professor, Tongji Hospital
Other Study IDs: CHALLENGE-03
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Liver Cancer; Emotional Disorder
MeSH Terms: conditions — Liver Neoplasms | interventions — Lysholm Knee Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Advanced unresectable HCC cohort: Cohort 1: Impact of ED on first-line therapy for advanced, unresectable HCC (n=243)
  Interventions: Other: Scale score
- Advanced unresectable ICC cohort: Cohort 2: Impact of ED on first-line therapy for advanced, unresectable intrahepatic cholangiocarcinoma (ICC) (n=175)
  Interventions: Other: Scale score
- Resectable high-risk HCC cohort: Cohort 3: Impact of ED on postoperative recurrence in resectable high-risk HCC (n=233)
  Interventions: Other: Scale score

INTERVENTIONS:
Other: Scale score — * The PHQ-9 rating scale and GAD-7 rating scale were used to screen for depression and anxiety symptoms in cancer patients;
    * The PSQI was used to assess the sleep quality index of cancer patients; ③ The PHQ-9 rating scale and GAD-7 rating scale were used to evaluate the depression and anxiety status of patient caregivers; ④ The European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) was used to assess the quality of life of cancer patients.

SUMMARY:
Hepatocellular carcinoma (HCC) carries a poor prognosis, with limited efficacy from current therapies including immune checkpoint inhibitors (ICIs). Concurrently, emotional distress (ED) is highly prevalent in cancer patients and is implicated in tumor progression via neuroendocrine-immune axis dysregulation (e.g., HPA axis activation, immunosuppressive TME). Emerging evidence, particularly from lung cancer, suggests ED may adversely impact ICI efficacy. However, its specific role and clinical significance in HCC, especially regarding ICI response, remain poorly understood.

To address this gap, we propose a large-scale, prospective, multicenter, multi-cohort study to systematically evaluate the impact of ED on treatment outcomes in HCC patients receiving immunotherapy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) carries a poor prognosis, with limited efficacy from current therapies including immune checkpoint inhibitors (ICIs). Concurrently, emotional distress (ED) is highly prevalent in cancer patients and is implicated in tumor progression via neuroendocrine-immune axis dysregulation (e.g., HPA axis activation, immunosuppressive TME). Emerging evidence, particularly from lung cancer, suggests ED may adversely impact ICI efficacy. However, its specific role and clinical significance in HCC, especially regarding ICI response, remain poorly understood.

To address this gap, we propose a large-scale, prospective, multicenter, multi-cohort study to systematically evaluate the impact of ED on treatment outcomes in HCC patients receiving immunotherapy.

This multi-cohort study comprises three independent cohorts:

Cohort 1: Impact of ED on first-line therapy for advanced, unresectable HCC (n=243).

In the recently published LEAP-012 study, the median progression-free survival (PFS) for advanced HCC receiving first-line transarterial chemoembolization (TACE) combined with immunotherapy and targeted therapy was 14.6 months. Based on an observed median PFS of 14.6 months for the overall population, a hazard ratio (HR) for tumor progression of approximately 1.7 for the ED group, and an estimated ED prevalence of 48.89%, we assumed exponential survival distributions for both groups. The overall survival function was constructed as:

S(t) = 0.4889 × exp(-1.7λ₀t) + 0.5111 × exp(-λ₀t) where λ₀ is the hazard rate for the non-ED group. Solving the key equation S(14.6)=0.5 numerically yields λ₀ ≈ 0.0357 per month. Consequently: Median PFS for the non-ED group = ln(2)/λ₀ ≈ 19.4 months Median PFS for the ED group = 19.4 / 1.7 ≈ 11.2 months With a two-sided alpha of 0.05, power (1-β) of 0.8, an accrual period of 12 months, and a maximum follow-up of 18 months, analysis using PASS 15 software indicated a required sample size of 194 subjects. Accounting for an estimated 20% dropout rate, a total of 243 participants will be enrolled.

Cohort 2: Impact of ED on first-line therapy for advanced, unresectable intrahepatic cholangiocarcinoma (ICC) (n=175).

In the TOPAZ-1 study, the median PFS for advanced biliary tract cancer receiving first-line chemotherapy combined with durvalumab was 12.9 months. Using the same calculation method as for Cohort 1, the estimated median PFS is approximately 9.8 months for the ED group and 17.0 months for the non-ED group. Considering the lower incidence of ICC, a longer accrual period is required. With a two-sided alpha of 0.05, power of 0.8, an accrual period of 24 months, and a maximum follow-up of 30 months, PASS 15 analysis indicated a required sample size of 140 subjects. Accounting for a 20% dropout rate, a total of 175 participants will be enrolled.

Cohort 3: Impact of ED on postoperative recurrence in resectable high-risk HCC (n=233).

In early-stage resectable HCC, patients with high-risk recurrence factors often experience early recurrence, with a reported median disease-free survival (DFS) of approximately 21.4 months. Using the same calculation method as for Cohort 1, the estimated median DFS is approximately 16.2 months for the ED group and 28.1 months for the non-ED group. With a two-sided alpha of 0.05, power of 0.8, an accrual period of 12 months, and a maximum follow-up of 24 months, PASS 15 analysis indicated a required sample size of 186 subjects. Accounting for a 20% dropout rate, a total of 233 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years, inclusive, regardless of gender.
* Presence of at least one radiologically measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (defined as a lesion with a longest diameter of ≥10 mm on CT scan).
* Newly diagnosed, treatment-naïve patients with hepatocellular carcinoma (HCC) or intrahepatic cholangiocarcinoma (ICC).
* Child-Pugh liver function score ≤ 7.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Absence of severe organic diseases affecting the heart, lungs, brain, or other major organs.

Exclusion Criteria:

* History of other malignancies.
* Recurrent HCC.
* Prior systemic therapy for HCC.
* Hepatic decompensation.
* History of severe psychiatric disorders.
* Current use of antidepressant or anxiolytic medication.
* Inability to comprehend or complete the assessment questionnaires.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult patients with newly diagnosed, treatment-naïve, unresectable HCC or ICC who are scheduled to receive guideline-recommended first-line immunotherapy-based regimens. Eligible participants must have at least one radiologically measurable lesion per RECIST 1.1 criteria, preserved liver function, and a good performance status. This population is designed to evaluate the impact of baseline emotional distress on immunotherapy outcomes in a representative cohort of patients with primary liver cancer initiating standard-of-care treatment.
Sampling Method: Probability Sample
Enrollment: 651 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | From date of enrollment until the date of first progress or date of death from any cause, whichever came first, assessed up to 60 months.
  In the three cohorts, PFS following immunotherapy was compared between primary liver cancer patients with and without emotional disorders.

SECONDARY OUTCOMES:
Overall survival(OS) | From date of enrollment until the date of death from any cause, assessed up to 96 months.
  In the three cohorts, OS following immunotherapy was compared between primary liver cancer patients with and without emotional disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Hepato-Pancreato-Biliary Surgery, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China